CLINICAL TRIAL: NCT02296203
Title: A PHASE II SINGLE-ARM STUDY OF CETUXIMAB PLUS IRINOTECAN AS RECHALLENGE 3RD-LINE TREATMENT OF KRAS, NRAS AND BRAF WILD-TYPE IRINOTECAN-PRETREATED METASTATIC COLORECTAL CANCER PATIENTS PROGRESSING AFTER AN INITIAL RESPONSE TO A 1ST-LINE CETUXIMAB-CONTAINING THERAPY AND A STANDARD 2ND-LINE
Brief Title: Cetuximab Rechallenge in Irinotecan-pretreated mCRC, KRAS, NRAS and BRAF Wild-type Treated in 1st Line With Anti-EGFR Therapy (CRICKET).
Acronym: CRICKET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GONO 10
Record Dates: First submitted 2014-10-15; First posted 2014-11-20 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: cetuximab rechallenge
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan

ARMS (1):
- cetuximab and irinotecan (Experimental)
  Interventions: Drug: cetuximab; Drug: irinotecan

INTERVENTIONS:
Drug: cetuximab
Drug: irinotecan

SUMMARY:
This is a multicentric, phase II single-arm study in which KRAS, NRAS and BRAF wild-type, irinotecan-resistant metastatic colorectal cancer patients progressing after an initial response to a first-line cetuximab-containing therapy, receive a rechallenge third-line treatment with cetuximab plus irinotecan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of colorectal adenocarcinoma;
* RAS and BRAF wild-type status;
* First-line irinotecan-based (FOLFIRI or FOLFOXIRI) cetuximab-containing therapy producing at least a partial response;
* First-line progression-free survival in response to cetuximab-containing therapy ≥6 months;
* Documentation of progression to first-line cetuximab within 4 weeks after last cetuximab administration;
* Time between the end of first-line therapy and the start of third-line treatment with cetuximab plus irinotecan ≥4 months;
* Second-line oxaliplatin-based (FOLFOXIRI, FOLFOX or XELOX) bevacizumab-containing therapy;
* Documentation of progression to second-line treatment;
* Measurable disease according to RECIST criteria v1.1;
* Have tumor tissue (of primary tumor and metastases or at least one of the two) available for biomarker analysis;
* Male or female patients > 18 years of age;
* ECOG Performance Status ≤ 2;
* Life expectancy of at least 3 months;
* Adequate bone marrow, liver and renal function assessed within 14 days before starting study treatment;
* Women of childbearing potential must have a negative blood pregnancy test at the baseline visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 months, are surgically sterile or are sexually inactive;
* Subjects and their partners must be willing to avoid pregnancy during the trial and until 6 months after the last trial treatment. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception as approved by the investigator, such as a two-barrier method or one-barrier method with spermicidal or intrauterine device. This requirement begins 2 weeks before receiving the first trial treatment and ends 6 months after receiving the last treatment;
* Signed informed consent obtained before any study specific procedure.

Exclusion Criteria:

* Active uncontrolled infections or active disseminated intravascular coagulation;
* Past or current history of malignancies other than colorectal carcinoma, except for curatively treated basal and squamous cell carcinoma of the skin cancer or in situ carcinoma of the cervix;
* Fertile women (< 12 months after last menstruation) and men of childbearing potential not willing to use effective means of contraception
* Women who are pregnant or are breastfeeding;
* Previous grade 3/4 infusion related reaction to cetuximab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-10; Primary Completion 2017-06-19 (Actual); Study Completion 2018-06-15 (Estimated)

PRIMARY OUTCOMES:
percentage of patients achieving a decrease equal or more than 30% in the sum of the longest diameters of target lesions | evaluation every 8 weeks until 48 weeks
  ORR is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria. The determination of clinical response will be based on investigator-reported measurements. Responses will be evaluated with a chest and abdominal computed tomography (CT) scan every 8 weeks. Patients who do not have an on-study assessment will be included in the analysis as non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Falcone, MD, PhD, Principal Investigator — U.O. Oncologia Medica 2 Universitaria, Università di Pisa - AOUP, Polo Oncologico, Area Vasta Nord-Ovest, Istituto Toscano Tumori
Locations (9):
- Italy (9):
  - AUSL DI FROSINONE - FROSINONE (FR) ONCOLOGIA MEDICA U.O. Oncologia Medica, Frosinone
  - Irccs Istituto Oncologico Veneto (Iov) - Padova (Pd) Oncologia Medica, Padua
  - Azienda Ospedaliero Universitaria Di Parma - U.O.Oncologia Medica, Parma
  - A.O. Universitaria Pisana - Pisa (Pi) Oncologia Medica, Pisa
  - AUSL 5 DI PISA - PISA (PI) ONCOLOGIA MEDICA oncologia medica Osp Lotti Pontedera, Pontedera
  - Ospedale Fatebenefratelli, Roma
  - Azienda Policlinico Umberto I - Oncologia Medica, Roma
  - Campus Biomedico, Roma
  - A.O. Universitaria S.Maria Della Misericordia Di Udine, Udine

REFERENCES:
- [Derived] Ciardiello D, Martinelli E, Troiani T, Mauri G, Rossini D, Martini G, Napolitano S, Famiglietti V, Del Tufo S, Masi G, Santini D, Avallone A, Pietrantonio F, Lonardi S, Di Maio M, Zampino MG, Fazio N, Bardelli A, Siena S, Cremolini C, Sartore-Bianchi A, Ciardiello F. Anti-EGFR Rechallenge in Patients With Refractory ctDNA RAS/BRAF wt Metastatic Colorectal Cancer: A Nonrandomized Controlled Trial. JAMA Netw Open. 2024 Apr 1;7(4):e245635. doi: 10.1001/jamanetworkopen.2024.5635. PMID 38592721
- [Derived] Martini G, Ciardiello D, Famiglietti V, Rossini D, Antoniotti C, Troiani T, Napolitano S, Esposito L, Latiano TP, Maiello E, Del Re M, Lonardi S, Aprile G, Santini D, Masi G, Avallone A, Normanno N, Pietrantonio F, Pinto C, Ciardiello F, Cremolini C, Martinelli E. Cetuximab as third-line rechallenge plus either irinotecan or avelumab is an effective treatment in metastatic colorectal cancer patients with baseline plasma RAS/BRAF wild-type circulating tumor DNA: Individual patient data pooled analysis of CRICKET and CAVE trials. Cancer Med. 2023 Apr;12(8):9392-9400. doi: 10.1002/cam4.5699. Epub 2023 Mar 7. PMID 36880426
- [Derived] Cremolini C, Rossini D, Dell'Aquila E, Lonardi S, Conca E, Del Re M, Busico A, Pietrantonio F, Danesi R, Aprile G, Tamburini E, Barone C, Masi G, Pantano F, Pucci F, Corsi DC, Pella N, Bergamo F, Rofi E, Barbara C, Falcone A, Santini D. Rechallenge for Patients With RAS and BRAF Wild-Type Metastatic Colorectal Cancer With Acquired Resistance to First-line Cetuximab and Irinotecan: A Phase 2 Single-Arm Clinical Trial. JAMA Oncol. 2019 Mar 1;5(3):343-350. doi: 10.1001/jamaoncol.2018.5080. PMID 30476968